CLINICAL TRIAL: NCT04618341
Title: A Clinical Study of Online Active Play Program With Adolescents During COVID-19 Lockdown
Brief Title: A Clinical Study of Online Active Play Program With Adolescents
Status: Completed | Type: Observational
Sponsor: Revival Active (Other)
Collaborators: L.E.A.D (Unknown); Aarogyam UK (Other)
Responsible Party: Sponsor
Other Study IDs: RAP/003
Record Dates: First submitted 2020-10-28; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Anxiety; Depression
Keywords: Adolescents; Online Active Revival Program
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the efficacy of an online, active play program (Revival Active Program) in reducing the symptoms of anxiety and depression in community-based adolescents,, a retrospective community based participatory research was conducted with 32 adolescents aged between 11-17 years old.

Program was conducted during Covid-19 lockdown from March 2020 to June 2020 to support children and families in isolation.

ELIGIBILITY:
Inclusion Criteria:

* Children at the online program for whole duration
* indicating a symptom level of, at minimum, above mean on anxiety and/or depression on self-report measures
* Parental consent before stating the program

Exclusion Criteria:

* Children at normal levels of mental health screening
* Children who did not complete the intervention period

Ages: 11 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Children who has attended online Revival Active Program (RAP) during COVID-19 lockdown
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Anxiety | Change from baseline anxiety at 6 weeks
  Screen for Child Anxiety Related Disorders (SCARED) child version was used to assess anxiety levels.
Depression | Change from baseline depression at 6 weeks
  Severity Measure for Depression child version was used to measure depression levels

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Patel, Study Director — Revival Active Limited; Tejal Patel, Study Director — Revival Active Limited; Nagamani Krishnamurthy, Principal Investigator — Aarogyam UK
Locations (1):
- Revival Active, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided